CLINICAL TRIAL: NCT07009184
Title: TGW211 for Click-Cleavable Imaging in HER2-Positive Cancers, a Phase 0/I Study.
Brief Title: TGW211 for Click-Cleavable Imaging in HER2-Positive Cancers.
Acronym: CleavHER
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Tagworks Pharmaceuticals BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 116650; 2025-520673-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: HER2 Positive Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Click-chemistry using [111In]In-DOTA-TCO-trastuzumab and trigger component TRG001 (TGW211) (Experimental): The goal and main intervention are to demonstrate safety and tolerability of click-chemistry using the intravenously administered radiolabeled (Indium-111) imaging tracer [111In]In-DOTA-TCO-trastuzumab in combination with an intravenously injected trigger component (TRG001). Following a cold pre dose trastuzumab to minimize antibody-sink effect, a radioactivity dose of 150 ± 20% MBq [111In]In-DOTA-TCO-trastuzumab is administered using a fixed microdose of protein up to 4.5 mg (< 30 nM). This is followed by intravenous administration of TRG001 in escalating dose levels. TRG001 cleaves [111In]In-DOTA-TCO-trastuzumab at the TCO-linker level. In subsequent cohorts the TRG001 dose level is escalated using a traditional 3+3 dose escalation design (38). After cleavage, the [111In]In-DOTA fragment is excreted via the urine.
  Interventions: Drug: [111In]In-DOTA-TCO-trastuzumab; Drug: Small molecule tetrazine trigger component

INTERVENTIONS:
Drug: [111In]In-DOTA-TCO-trastuzumab — [111In]In-DOTA-TCO-trastuzumab is a chemically cleavable [111In]In-labeled trastuzumab conjugate that is administered first to the patient, it accumulates in HER2-positive tumors and internalizes in HER2-expressing tumor cells.
Drug: Small molecule tetrazine trigger component — TRG001 is a small molecule tetrazine trigger that reacts with [111In]In-TGW211-DC in blood and extracellular space thus releasing a fast clearing [111In]In-DOTA containing fragment which is rapidly eliminated via the kidney. Because of its non-cell permeable nature, TRG001 does not reach [111In]In-TGW211-DC inside tumor cells and therefore the radioactivity inside tumor cells is retained by the tumor.

SUMMARY:
In recent years, there is increasing interest in antibodies for imaging, antibody-drug conjugates (ADC) and targeted radionuclide therapy (TRT). With these techniques, antibodies are used as a vector to deliver a cytotoxic drug or radionuclide for therapy or nuclear medicine imaging. One such antibody-based vector suitable for delivering a cytotoxic drug or radionuclide is trastuzumab, which targets HER2 that is overexpressed in cancers such as breast, gastric and gastroesophageal junction carcinomas. Unfortunately, antibodies generally have a very long circulation time (>20-30 days) that often result in unfavorable background noise in the healthy organs in imaging or toxicity when trastuzumab is bound to a therapeutic radionuclide for radioimmunotherapy. There is thus a need to increase the speed of excretion of antibodies or release the antibody from its payload. Ideally, the clinician would like to appropriately time the elimination of radioactivity to achieve an optimal tumor to non-tumor ratio. To this aim, Tagworks Pharmaceuticals developed a new class of chemically cleavable radiolabeled conjugates that release the radiolabel on demand upon reaction with a small molecule "the trigger" (TRG001).

DETAILED DESCRIPTION:
In the last decade, there was increasing interest in antibody mediated imaging, ADCs, and TRT. There are now antibodies targeting human epidermal growth factor receptor (HER2), trophoblast antigen 2 (TROP2), nectin-4, folate receptor alpha, prostate-specific membrane antigen (PSMA), among others. These drugs use antibodies as a vector to deliver a (cytotoxic) payload for imaging or therapeutic purposes. After binding to the receptor, the antibody-based therapy is internalized and introduces the drug or radionuclide to the inside of the (cancer) cell. This causes the cell to die or light up, driven by the radionuclide of choice.

One of the most used antibodies in the clinic, is trastuzumab. Trastuzumab (Herceptin®) is a recombinant humanized IgG1 monoclonal antibody directed against the HER2 receptor. HER2 is a member of the epidermal growth factor receptor (EGFR) family of receptor tyrosine kinase, and its expression is upregulated in several tumor types. HER2 is a well-defined, clinically relevant internalizing tumor target expressed at high levels in multiple different cancer types. Breast and gastric/gastroesophageal cancers have been the focus of HER2-targeted therapies, but HER2 overexpression occurs in various other malignancies of epithelial origin, such as, gastric, ovarian, bladder, salivary gland, endometrial, pancreatic, and non-small-cell lung cancer. Binding of trastuzumab to HER2-expressing cells suppresses HER2 signaling pathways, induces cell cycle arrest and mediates antibody-dependent cell-mediated cytotoxicity. Trastuzumab therapy can also be combined with chemotherapy to obtain synergistic effects, and to limit the often-observed resistance against the therapy. HER2 plays an important role in oncogenic transformation, oncogenesis, and metastatic spread of cancer. Overexpression is associated with a poor prognosis and predicts a poor response to several treatment modalities.

Molecular imaging techniques substitute for invasive biopsy procedures, exhibiting an immense advantage over other available markers. Nuclear imaging using radioactively labeled trastuzumab can easily distinguish patients who are responsive to HER2-targeted therapy from patients who are primarily resistant to anti-HER2 treatment. For this purpose, trastuzumab has been functionalized with chelators such as DOTA, EDTA and deferoxamine for radiolabeling with a variety of isotopes for nuclear medicine imaging. Trastuzumab can be labeled with Indium-111 (gamma decay) or Zirconium-89 (positron decay) to assess HER2-positive disease in patients using single photon emission computed tomography (SPECT) or positron emission tomography (PET), respectively.

Trastuzumab labeled with a therapeutic radionuclide could be an attractive alternative to antibody treatment or chemotherapy. A HER2-targeted antibody such as trastuzumab, labeled with therapeutic radionuclides (e.g., Lutetium-177, Yttrium-90, Actinium-225, Thorium-227, etc.) has the potential to markedly improve current HER2 targeted cancer therapy. The bystander effect (the killing of neighboring receptor-negative cancer cells by radiation crossfire) would be especially beneficial for the inherently heterogeneous metastatic tumors. In addition, contrary to standard HER2-targeted therapies, resistance to radiation is unlikely to occur. Trastuzumab-based radiotherapy has been tested in patients with trastuzumab radiolabeled with alpha-emitting Lead-212 (15) and beta-emitting Lutetium-177 and appeared to be safe.

A limitation of the use of monoclonal antibodies, such as trastuzumab, as vectors for radioactivity is their slow clearance rates and thus long blood circulation time (20). Sustained circulation increases the uptake in solid tumors making them useful as vectors, but also causes significant side effects to the healthy organs such as to the bone marrow, and liver. This is particularly applicable to radionuclide therapy as the range of alpha (e.g. Actinium-225) and beta (e.g. Lutetium-177) particles ranges from <0.4 to a few millimeters and causes serious damage to bone marrow cells resulting in severe, dose-limiting myelotoxicity for the patient, significantly limiting the therapeutic effect. This is one of the main reasons antibody-based radionuclide therapy never became a treatment for solid tumors. Moreover, the long circulation time of antibodies increases the time to image with [111In]In-trastuzumab SPECT or [89Zr]Zr-trastuzumab PET imaging to several days post tracer injection due to unfavorable background noise in the circulation and healthy organs. There is thus a need to increase the speed of excretion of antibodies or release the antibody from its (cytotoxic) payload. Ideally, the clinician would have complete temporal control over radioactivity clearance from circulation to achieve an optimal tumor to non-tumor ratio.

Click-chemistry is a relatively novel chemistry method for which the Nobel prize was awarded in 2022. One method to use click-chemistry is to create click-cleavable radiolabeled conjugates. This has the potential to significantly decrease the side effects associated with radiopharmaceuticals in cancer patients, thus increasing the therapeutic effect. Tagworks Pharmaceuticals, with their TGW211 program, is proposing the use of a new class of radiolabeled monoclonal antibodies where the radionuclide is bound to the antibody (trastuzumab in the current study) via a chemically cleavable trans-cyclooctene (TCO) linker which, upon click reaction with an exogenous small molecule tetrazine, "the trigger" (TRG001), releases a fragment containing the radiolabeled chelate ([111In]In-DOTA fragment) instantaneously and quantitatively. Upon release in the blood circulation, the cleaved radiolabeled fragment ([111In]In-DOTA) is rapidly eliminated via the urine, as shown previously for unmodified chelates, thereby rapidly decreasing systemic exposure to radioactivity. Trigger-mediated cleavage occurs only extracellularly and not inside tumor cells as the trigger is cell impermeable and is administered post administration of the radiolabeled conjugate, once it has been taken up by tumor cells. In this study, we will evaluate safety and assess the time window where cleavage should be done for an optimal tumor-to-healthy organ ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent and willing and able to comply with study requirements.
2. Male or Female aged ≥ 18 years.
3. Histologically confirmed HER2-positive cancer (IHC 3+ or IHC 2+ AND FISH+) with at least 1 measurable target lesion of at least 10 mm on CT or MRI based on RECIST v1.1, assessed by the investigator to enable adequate SPECT/CT imaging.
4. WHO performance status (ECOG) of 0 or 1.
5. Adequate organ and bone marrow function, evidenced by the following laboratory results:

   1. Absolute neutrophil count ≥ 1.5 x 10^9 /l;
   2. Platelet count ≥ 100 x 10^9 /l;
   3. Hemoglobin ≥ 9.0 g/dl or 5.6 mmol/l;
   4. Total bilirubin ≤ 1.5 x the upper limit of normal (ULN);
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN (or ≤ 5.0 x ULN in the presence of liver metastases);
   6. Serum creatinine ≤ 1.5 x ULN; - Estimated Glomerular Filtration Rate (eGFR)* ≥ 60 ml/min/1.73 m2 ; *preferably calculated with CKD-EPI formula.

Exclusion Criteria:

1. Medical history of myocardial infarction within 6 months before participation or symptomatic CHF (New York Heart Association Class III to IV).
2. QT interval corrected by Fridericia's formula (QTcF) ≥ 470 msec on screening ECG or congenital long QT syndrome.
3. Has a history of (non-infectious) ILD/pneumonitis that required steroids or has current or suspected ILD/pneumonitis.
4. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g, pulmonary embolism within 3 months of trial participation, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc.).
5. Has an uncontrolled infection requiring systemic antibiotics, antivirals, or antifungals.
6. Participation in another clinical study with an investigational product during the past 6 weeks.
7. Concurrent enrolment in another clinical study unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study.
8. Pregnant or breastfeeding women, where pregnancy is defined as the time between conception and termination of gestation, confirmed by a positive urinary or serum pregnancy test.
9. Women of childbearing potential (WOCBP), defined as women physiologically capable of becoming pregnant and no evidence of post-menopausal status, unless they use highly effective methods of contraception or abstain from sexual activity for 30 days after investigational drug administration. Male partners of female patients should also use a condom during intercourse for 30 days after investigational drug administration to the partner to prevent them from fathering a child.
10. Male patients in the reproductive age, not willing or able to use a condom or abstain from sexual activity for 30 days after investigational drug administration. WOCBP partners of sexually active male patients should also use a highly effective contraception method during intercourse for 30 days after investigational drug administration of the partner.
11. Known allergy or hypersensitivity to any of the investigational drugs or its excipients.
12. Any condition which, in the opinion of the investigator, would preclude participation in the study.
13. Second active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events using the CTCAE version 5.0. | From enrollment to end of treatment at 14 days after last dose of investigational product.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No